CLINICAL TRIAL: NCT03022032
Title: The HOPE Trial: Helping Our Patients Excel, and The SMART Study: Symptom Management and Reporting
Brief Title: The HOPE Trial and the SMART Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Alexi A. Wright, MD, Alexi. A Wright, MD, MPH, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-477; 1R21NR018532 (NIH)
Record Dates: First submitted 2017-01-06; First posted 2017-01-16 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Gynecologic Cancer
Keywords: Gynecologic cancer
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Comparing Steps Collected by Accelerometer (HOPE) (Experimental): * 10 patients will be enrolled in stage 1 to refine the HOPE App intervention
  * All participants will receive :
    * HOPE App
    * The Fitbit Zip
    * The Fitbit Charge 2 The amount of step collected by each device will be compared. This will allow the team to identify which wearable accelerometer to use in stage 2
  Interventions: Device: Fitbit Zip; Other: HOPE App; Device: Fitbit Charge 2
- Usual care (HOPE) (Other): Stage 2 will consist of arm 2-5 and will enroll 100 randomized patients.
  * Usual care
  * The app will also collect passive data from the smartphone
  Interventions: Other: HOPE App; Other: Standard of Care
- Wearable accelerometer (HOPE) (Experimental): * Participants will be asked to wear the Fitbit
  * The Hope App will measure daily steps
  * The app will also collect passive data from the smartphone
  Interventions: Other: HOPE App; Device: Fitbit Charge 2
- Refined smartphone app (HOPE) (Experimental): * Participants will be prompted to answer questions about their quality of life and physical health daily
  * The HOPE App will present tailored advice to improve symptoms if one or more low-risk toxicities are reported. If the symptoms are determined to be high-risk, the App will prompt the patient to call their clinician.
  * The app will also collect passive data from the smartphone
  Interventions: Other: HOPE App
- Refined smartphone app and accelerometer (HOPE) (Experimental): * Participants will be prompted to answer questions about their quality of life and physical health daily
  * The HOPE App will present tailored advice to improve symptoms if one or more low-risk toxicities are reported. If the symptoms are determined to be high-risk, the App will prompt the patient to call their clinician.
  Participants will be asked to wear the Fitbit
  -The Hope App will measure daily steps The app will also collect passive data from the smartphone
  Interventions: Other: HOPE App
- SMART Study Arm (Experimental): * Two smartphone apps and a wearable accelerometer (Fitbit) in 30 patients with gynecologic cancers receiving chemotherapy at two NCI Community Oncology sites.
  * The SMART intervention refers to the combination of both smartphone apps (SMART app and Beiwe app) and the accelerometer (Fitbit).
  * The SMART app is the technology that is actively collecting symptom reporting information from patients (e.g. patients are receiving surveys, recording their symptoms daily, and receiving tailored symptom management materials on their phone in response).
  * The Beiwe app is the technology involved in the passive data collection of participants' symptoms (GPS and accelerometer data) without their involvement.
  Interventions: Other: SMART Study Intervention

INTERVENTIONS:
Device: Fitbit Zip — Fitbit Zip
  Arms: Comparing Steps Collected by Accelerometer (HOPE)
Other: HOPE App — HOPE App
  Arms: Comparing Steps Collected by Accelerometer (HOPE); Refined smartphone app (HOPE); Refined smartphone app and accelerometer (HOPE); Usual care (HOPE); Wearable accelerometer (HOPE)
Other: Standard of Care — Standard of Care
  Arms: Usual care (HOPE)
Device: Fitbit Charge 2 — Fitbit Charge 2
  Arms: Comparing Steps Collected by Accelerometer (HOPE); Wearable accelerometer (HOPE)
Other: SMART Study Intervention — SMART study app + Beiwe study app + Fitbit
  Arms: SMART Study Arm

SUMMARY:
This research study is evaluating a new smartphone application named the "Helping Our Patients Excel (HOPE)" app with a Fitbit device. The SMART Study is a sub-study of the HOPE Trial. Both studies evaluate an almost identical intervention using a Fitbit device and smartphone app(s) with the goal of improving quality-of-life for women with gynecologic cancers.

DETAILED DESCRIPTION:
The HOPE Trial:

The first goal of this study is to adapt and refine an existing smartphone app, paired with a wearable accelerometer, to assess patients' symptoms in a population of patients with gynecologic cancers receiving palliative chemotherapy. An existing app will be customized to collect patient-reported toxicities using the Patient-Reported Outcome (PRO) version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) and offer patients feedback about how to manage their symptoms. Patient symptoms will be risk-stratified. Patients with low-risk toxicities (grades 1 & 2) will receive tailored educational information, while patients with serious toxicities (grades 3 & 4) will receive alerts to call their clinician. In the first phase of the study, we will conduct an initial assessment of the app with a diverse group of 10 patients to refine the app and test two different wearable accelerometers (i.e. Fitbit Zip and Fitbit Charge 2) before pilot testing.

The second goal of this study is to conduct a pilot randomized controlled trial (RCT) of the smartphone app and/or wearable accelerometer (i.e. Fitbit Zip or Fitbit Charge 2) to assess the feasibility, acceptability, and preliminary efficacy of our intervention. During the second phase of the study, we will conduct a 4-arm pilot RCT in 100 patients with gynecologic cancers receiving palliative chemotherapy to establish preliminary effect sizes. Participants will be randomized to: 1) Fitbit+active app, 2) Fitbit+passive app, 3) Active app, or 4) Passive app.

We expect that the results of this pilot RCT, which is supported by the National Cancer Institute, National Palliative Care Research Center, and the Dana-Farber Cancer Institute Department of Medical Oncology, will provide a low-cost, scalable system to assess patients' symptoms, address low-risk toxicities, and alert clinicians when patients have toxicities that require intervention with the goal of reducing patient suffering and the use of high-intensity, hospital-based health care.

The SMART Study:

The overall goals of this study are to test the combination of two smartphone research platforms and a wearable accelerometer for use in NCI Community Oncology Research Program (NCORP) sites to improve cancer patients' quality of life and symptom management. The SMART Study (Symptom Management and Reporting Toxicities) has a single-arm research design and aims to assess the feasibility, acceptability, and perceived efficacy of a wearable accelerometer and two smartphone apps in 30 patients receiving chemotherapy to treat recurrent gynecologic cancers.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years of age
* Who plan to receive chemotherapy at DFCI to treat recurrent, incurable gynecologic cancers (ovarian, uterine, cervical) that have recurred despite ≥1 prior treatments.
* Own a smart-phone (Android or iOS)
* Capable of downloading and running the study app without assistance
* Can read and provide informed consent in English
* Do not have cognitive or visual impairments that would preclude use of the app.

Exclusion Criteria:

* Patients will be ineligible if they are participating in an investigational drug treatment trial that requires structured symptom or toxicity reporting at the time of enrollment.
* Patients with severe cognitively impairments
* Who appear too weak
* Emotionally distraught
* Agitated or ill to participate, as judged by either the research study staff or an oncology provider, will be excluded.
* Patients who are unable to provide informed consent in English will be excluded because the smartphone app intervention is only available in English at this time.
* Children and young adults up to age 18 will be excluded because the diagnosis of metastatic gynecologic cancers in this age group is rare and the proposed instruments are not designed for people of those ages.
* Patients with a life expectancy of ≤6 months, as determined by their oncology providers, will be excluded since they cannot participate in all of the required data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexi A Wright, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HOPE Pre-Pilot: 10 patients will be enrolled in stage 1 to refine the HOPE App intervention. All participants will receive the HOPE App and The Fitbit Zip or The Fitbit Charge 2. This will allow the team to identify which wearable accelerometer to use in stage 2.
- Refined Smartphone App and Accelerometer (HOPE): Participants received the FitBit Charge 2 and access to the HOPE smartphone app. The HOPE app presented tailored advice if one or more low-risk symptoms were reported and prompted the patient to call their clinician for high-risk symptoms.
- Wearable Accelerometer (HOPE): Participants were asked to wear the Fitbit Charge 2. The HOPE app will also collect passive smartphone data.
- Refined Smartphone App (HOPE): Participants received access to the HOPE smartphone app. The HOPE app presented tailored advice if one or more low-risk symptoms were reported and prompted the patient to call their clinician for high-risk symptoms.
- Usual Care (HOPE): The HOPE app will collect passive data from the smartphone.
- SMART Study Arm: Participants received the Fitbit Charge 2 and access to the smartphone app. The app presented tailored advice if one or more low-risk symptoms were reported and prompted the patient to call their clinician for high-risk symptoms.
Period: Overall Study
Arm/Group | HOPE Pre-Pilot | Refined Smartphone App and Accelerometer (HOPE) | Wearable Accelerometer (HOPE) | Refined Smartphone App (HOPE) | Usual Care (HOPE) | SMART Study Arm
Started | 10 | 23 | 21 | 22 | 22 | 4
Completed | 10 | 23 | 21 | 22 | 22 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Comparing Steps Collected by Accelerometer (HOPE): * 10 patients will be enrolled in stage 1 to refine the HOPE App intervention
  * All participants will receive :
    * HOPE App
    * The Fitbit Zip
    * The Fitbit Charge 2 The amount of step collected by each device will be compared. This will allow the team to identify which wearable accelerometer to use in stage 2
  Fitbit Zip: Fitbit Zip
  HOPE App: HOPE App
  Fitbit Charge 2: Fitbit Charge 2
- Refined Smartphone App and Accelerometer (HOPE): * Participants will be prompted to answer questions about their quality of life and physical health daily
  * The HOPE App will present tailored advice to improve symptoms if one or more low-risk toxicities are reported. If the symptoms are determined to be high-risk, the App will prompt the patient to call their clinician.
  Participants will be asked to wear the Fitbit
  -The Hope App will measure daily steps The app will also collect passive data from the smartphone
  HOPE App: HOPE App
- Wearable Accelerometer (HOPE): * Participants will be asked to wear the Fitbit
  * The Hope App will measure daily steps
  * The app will also collect passive data from the smartphone
  HOPE App: HOPE App
  Fitbit Charge 2: Fitbit Charge 2
- Refined Smartphone App (HOPE): * Participants will be prompted to answer questions about their quality of life and physical health daily
  * The HOPE App will present tailored advice to improve symptoms if one or more low-risk toxicities are reported. If the symptoms are determined to be high-risk, the App will prompt the patient to call their clinician.
  * The app will also collect passive data from the smartphone
  HOPE App: HOPE App
- Usual Care (HOPE): Stage 2 will consist of arm 2-5 and will enroll 100 randomized patients.
  * Usual care
  * The app will also collect passive data from the smartphone
  HOPE App: HOPE App
  Standard of Care: Standard of Care
- SMART Study Arm: * Two smartphone apps and a wearable accelerometer (Fitbit) in 30 patients with gynecologic cancers receiving chemotherapy at two NCI Community Oncology sites.
  * The SMART intervention refers to the combination of both smartphone apps (SMART app and Beiwe app) and the accelerometer (Fitbit).
  * The SMART app is the technology that is actively collecting symptom reporting information from patients (e.g. patients are receiving surveys, recording their symptoms daily, and receiving tailored symptom management materials on their phone in response).
  * The Beiwe app is the technology involved in the passive data collection of participants' symptoms (GPS and accelerometer data) without their involvement.
  SMART Study Intervention: SMART study app + Beiwe study app + Fitbit
- Total: Total of all reporting groups
Arm/Group | Comparing Steps Collected by Accelerometer (HOPE) | Refined Smartphone App and Accelerometer (HOPE) | Wearable Accelerometer (HOPE) | Refined Smartphone App (HOPE) | Usual Care (HOPE) | SMART Study Arm | Total
Number analyzed (Participants) | 10 | 23 | 21 | 22 | 22 | 4 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.29) | 61.52 (13.36) | 63.76 (8.43) | 62.09 (8.19) | 59.64 (9.31) | 65.50 (8.85) | 60.75 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 23 | 21 | 22 | 22 | 4 | 102
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 10 | 22 | 21 | 22 | 21 | 3 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Marital Status [Count of Participants; unit: Participants]
  Married | 8 | 14 | 12 | 14 | 14 | 2 | 64
  Divorced/Separated | 0 | 5 | 3 | 2 | 3 | 2 | 15
  Never Married | 1 | 3 | 4 | 2 | 4 | 0 | 14
  Widowed | 1 | 1 | 2 | 2 | 1 | 0 | 7
  Missing | 0 | 0 | 0 | 2 | 0 | 0 | 2
Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 3 | 0 | 1 | 0 | 5
  Black or African American | 2 | 1 | 1 | 0 | 3 | 0 | 7
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 20 | 15 | 21 | 17 | 4 | 83
  Other | 1 | 0 | 1 | 1 | 1 | 0 | 4
  Don't know | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Refuse to answer | 1 | 0 | 0 | 0 | 0 | 0 | 1
Last grade level completed [Count of Participants; unit: Participants]
  8th grade or less | 0 | 0 | 0 | 0 | 0 | 0 | 0
  9 - 11th grade | 1 | 0 | 0 | 0 | 0 | 0 | 1
  High school graduate or GED | 0 | 3 | 0 | 3 | 2 | 1 | 9
  Vocational or Technical training | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Associate degree or some college | 3 | 5 | 5 | 6 | 5 | 1 | 25
  Bachelor's degree | 0 | 5 | 9 | 3 | 8 | 2 | 27
  Advanced degree | 6 | 10 | 5 | 10 | 7 | 0 | 38
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Don't know | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Refused | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility (≥60% Enrollment Rate of Eligible Patients; ≥70% Survey Adherence; ≥80% FitBit Adherence) and Acceptability (≥60% Would Recommend the Intervention; <30% Rate the Study as Burdensome/Wish They Had Not Participated) in HOPE Pre-Pilot (n=10)
Description: This outcome was limited to the HOPE pre-pilot, consisting of 10 patients. This open pilot aimed to identify patient preference of Fitbit Zip or Fitbit Charge 2 and whether this study was burdensome. This outcome informed appropriate study procedures before launching to a larger study with four arms across multiple sites.
  Feasibility defined as (1) greater than or equal to 60% enrollment rate among eligible patients approached, (2) greater than or equal to 70% adherence to daily smartphone surveys, (3) greater than or equal to 80% adherence to Fitbits at least 4 days per week. Acceptability defined as responses to 3 questions: (1) "Participating in this study placed a substantial burden on me." (2) "I wish I had not agreed to participate in this study." and (3) "I would recommend the application to a friend going through treatment."
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | HOPE Pre-pilot
Number analyzed (Participants) | 10
Participants
  Feasibility - (1) greater than or equal to 60% enrollment rate among eligible patients approached | 10
  Feasibility - (2) greater than or equal to 70% adherence to daily smartphone surveys | 7
  Feasibility - (3) greater than or equal to 80% adherence to Fitbits at least 4 days per week | 9
  Acceptability - (1) "Participating in this study placed a substantial burden on me." | 1
  Acceptability - (2) "I wish I had not agreed to participate in this study." | 1

2. Primary Outcome: Number of Participants Who Preferred the FitBit Zip vs. Number of Participants Who Preferred the FitBit Charge HR in the HOPE Pre-Pilot Study (n=10)
Description: This outcome was limited to the HOPE Pre-pilot, consisting of 10 patients. This open pilot aimed to identify patient preference of Fitbit Zip or Fitbit Charge 2 and whether this study was burdensome. This outcome informed appropriate study procedures before launching to a larger study with four arms across multiple sites.
  This outcome is participant preference of the Fitbit Zip vs. Fitbit Charge in the HOPE Pre-Pilot study.
Time Frame: 30 days
Population: This outcome was limited to the HOPE pilot, consisting of 10 patients.
Measure: Number; unit: participants
Groups:
- HOPE Pre-pilot: Single arm pre-pilot of 10 participants.
Arm/Group | HOPE Pre-pilot
Number analyzed (Participants) | 10
participants
  Preferred FitBit Charge | 9
  Preferred FitBit Zip | 1

3. Primary Outcome: Feasibility (i.e. ≥50% 3-month Adherence Rates to Both Smartphone Apps and the Wearable Accelerometer) in the SMART Study
Description: SMART Study: Participants received the Fitbit Charge 2 and access to the smartphone app. The app presented tailored advice if one or more low-risk symptoms were reported and prompted the patient to call their clinician for high-risk symptoms.
  Feasibility will be defined as greater than or equal to 50% 3-month adherence rates to both smartphone apps and the wearable accelerometer.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Groups:
- SMART Study: Single arm pre-pilot feasibility and acceptability testing of SMART at University of New Mexico and Sanford Health (Sioux Falls, South Dakota).
Arm/Group | SMART Study
Number analyzed (Participants) | 4
Participants | 4

4. Primary Outcome: Acceptability (i.e. ≥60% of Study Participants Would Recommend the Intervention to Other Patients; and <30% of Patients Rate the Study as Burdensome or Wish They Had Not Participated) in the SMART Study
Description: SMART Study: Participants received the Fitbit Charge 2 and access to the smartphone app. The app presented tailored advice if one or more low-risk symptoms were reported and prompted the patient to call their clinician for high-risk symptoms.
  Acceptability defined as responses to three questions: (1) "Participating in this study placed a substantial burden on me."; (2) "I wish I had not agreed to participate in this study."; and (3) "I would recommend the application to a friend going through treatment."
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | SMART Study
Number analyzed (Participants) | 4
Participants
  Acceptability - (1) "Participating in this study placed a substantial burden on me." | 0
  Acceptability - (2) "I wish I had not agreed to participate in this study." | 0
  Acceptability - (3) "I would recommend the application to a friend going through treatment." | 4

5. Secondary Outcome: Anxiety as Assessed by GAD-7 (HOPE RCT)
Description: Patients' GAD-7 measurements taken at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. [The General Anxiety Disorder-7 (GAD-7) total score has a minimum value of 0 and a maximum value of 21, with higher values corresponding to worse outcome.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: GAD-7 Total score
Groups:
- Arm 1: Fitbit + Active App: Participants received the Fitbit Charge 2 and access to the HOPE smartphone app. The HOPE app presented tailored advice if one or more low-risk symptoms were reported and prompted the patient to call their clinician for high-risk symptoms.
- Arm 2: Fitbit+Passive App: Participants were asked to wear the Fitbit Charge 2. The HOPE app will also collect passive smartphone data.
- Arm 3: Active App: Participants received access to the HOPE smartphone app. The HOPE app presented tailored advice if one or more low-risk symptoms were reported and prompted the patient to call their clinician for high-risk symptoms
- Arm 4: Passive App: The HOPE app will collect passive data from the smartphone.
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit+Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
GAD-7 Total score
  Baseline: number analyzed (Participants) | 23 | 19 | 22 | 20
  Baseline | 3.43 (2.98) | 3.74 (4.19) | 5.45 (4.82) | 4.10 (3.43)
  30 days post-baseline: number analyzed (Participants) | 12 | 11 | 11 | 15
  30 days post-baseline | 3.17 (3.24) | 5.09 (4.46) | 2.64 (2.54) | 4.00 (2.24)
  90 days post-baseline: number analyzed (Participants) | 8 | 8 | 13 | 14
  90 days post-baseline | 3.50 (3.55) | 3.38 (4.03) | 2.92 (2.47) | 3.07 (2.13)
  180 days post-baseline: number analyzed (Participants) | 9 | 9 | 12 | 9
  180 days post-baseline | 0.78 (0.97) | 3.78 (4.09) | 3.00 (2.26) | 3.22 (2.82)

6. Secondary Outcome: Depression as Assessed by PHQ-9 (HOPE RCT)
Description: Patients' PHQ-9 measurements taken at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {The Patient Health Questionnaire (PHQ-9) total score has a minimum value of 0 and a maximum value of 27, with higher values corresponding to worse outcome.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: PHQ-9 total score
Groups:
- Arm 2: Fitbit + Passive App: Participants were asked to wear the Fitbit Charge 2. The HOPE app will also collect passive smartphone data.
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
PHQ-9 total score
  Baseline: number analyzed (Participants) | 23 | 20 | 22 | 22
  Baseline | 4.43 (3.73) | 3.70 (3.48) | 4.95 (3.61) | 5.59 (4.62)
  30 days post-baseline: number analyzed (Participants) | 10 | 12 | 11 | 15
  30 days post-baseline | 3.20 (4.18) | 4.58 (4.46) | 3.27 (2.90) | 4.80 (3.38)
  90 days post-baseline: number analyzed (Participants) | 10 | 12 | 13 | 15
  90 days post-baseline | 5.90 (4.95) | 4.58 (5.04) | 3.46 (3.26) | 3.87 (1.96)
  180 days post-baseline: number analyzed (Participants) | 9 | 9 | 12 | 11
  180 days post-baseline | 1.22 (1.39) | 3.56 (4.00) | 3.42 (2.43) | 5.09 (2.98)

7. Secondary Outcome: Patient Well-being as Assessed by FACIT-Pal (HOPE RCT)
Description: Patients' FACIT-Pal measurements taken at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {The Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-Pal) total score has a minimum value of 0 and a maximum value of 184, with higher values corresponding to better outcome.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Total score
  Baseline | 142.1 (24.3) | 147.0 (23.2) | 139.7 (22.4) | 139.4 (21.1)
  30 days post-baseline: number analyzed (Participants) | 12 | 13 | 11 | 15
  30 days post-baseline | 150.7 (22.0) | 145.7 (26.4) | 147.4 (19.6) | 145.6 (18.7)
  90 days post-baseline: number analyzed (Participants) | 10 | 13 | 13 | 15
  90 days post-baseline | 132.3 (27.2) | 143.8 (34.3) | 150.9 (20.1) | 141.0 (18.4)
  180 days post-baseline: number analyzed (Participants) | 9 | 10 | 12 | 11
  180 days post-baseline | 161.4 (15.6) | 155.2 (22.8) | 144.1 (17.7) | 140.4 (23.6)

8. Secondary Outcome: Constipation as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 1-3 constipation at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 23 | 21 | 21 | 22
  Baseline | 10 | 6 | 10 | 11
  30 days post-baseline: number analyzed (Participants) | 12 | 13 | 10 | 15
  30 days post-baseline | 5 | 2 | 5 | 8
  90 days post-baseline: number analyzed (Participants) | 10 | 13 | 12 | 15
  90 days post-baseline | 2 | 6 | 5 | 8
  180 days post-baseline: number analyzed (Participants) | 9 | 9 | 12 | 11
  180 days post-baseline | 4 | 6 | 8 | 7

9. Secondary Outcome: Diarrhea as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 1-3 diarrhea at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 23 | 20 | 22 | 22
  Baseline | 10 | 8 | 7 | 11
  30 days post-baseline: number analyzed (Participants) | 12 | 12 | 11 | 15
  30 days post-baseline | 5 | 3 | 4 | 5
  90 days post-baseline: number analyzed (Participants) | 10 | 12 | 13 | 15
  90 days post-baseline | 5 | 5 | 4 | 9
  180 days post-baseline: number analyzed (Participants) | 9 | 9 | 12 | 11
  180 days post-baseline | 0 | 2 | 2 | 4

10. Secondary Outcome: Nausea as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 1-3 nausea at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 23 | 20 | 22 | 22
  Baseline | 12 | 7 | 11 | 12
  30 days post-baseline: number analyzed (Participants) | 12 | 12 | 11 | 13
  30 days post-baseline | 7 | 4 | 5 | 7
  90 days post-baseline: number analyzed (Participants) | 10 | 12 | 13 | 14
  90 days post-baseline | 7 | 1 | 6 | 11
  180 days post-baseline: number analyzed (Participants) | 9 | 8 | 12 | 12
  180 days post-baseline | 2 | 1 | 5 | 8

11. Secondary Outcome: Vomiting as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 1-3 vomiting at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 22 | 20 | 22 | 22
  Baseline | 2 | 1 | 4 | 5
  30 days post-baseline: number analyzed (Participants) | 12 | 12 | 11 | 15
  30 days post-baseline | 2 | 0 | 2 | 1
  90 days post-baseline: number analyzed (Participants) | 9 | 11 | 13 | 15
  90 days post-baseline | 3 | 0 | 1 | 1
  180 days post-baseline: number analyzed (Participants) | 8 | 9 | 12 | 11
  180 days post-baseline | 1 | 1 | 3 | 3

12. Secondary Outcome: Numbness and Tingling as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 1-3 numbness and tingling at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 23 | 20 | 20 | 22
  Baseline | 10 | 14 | 11 | 15
  30 days post-baseline: number analyzed (Participants) | 12 | 12 | 10 | 15
  30 days post-baseline | 8 | 10 | 4 | 11
  90 days post-baseline: number analyzed (Participants) | 10 | 10 | 13 | 14
  90 days post-baseline | 6 | 7 | 7 | 11
  180 days post-baseline: number analyzed (Participants) | 9 | 9 | 11 | 11
  180 days post-baseline | 5 | 7 | 4 | 5

13. Secondary Outcome: Dizziness as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 1-3 dizziness at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 23 | 19 | 21 | 22
  Baseline | 6 | 5 | 3 | 7
  30 days post-baseline: number analyzed (Participants) | 12 | 12 | 10 | 15
  30 days post-baseline | 5 | 0 | 2 | 2
  90 days post-baseline: number analyzed (Participants) | 10 | 14 | 13 | 15
  90 days post-baseline | 4 | 2 | 2 | 1
  180 days post-baseline: number analyzed (Participants) | 9 | 9 | 11 | 11
  180 days post-baseline | 1 | 1 | 1 | 4

14. Secondary Outcome: Abdominal Pain as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 1-3 abdominal pain at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 23 | 20 | 22 | 22
  Baseline | 12 | 8 | 10 | 16
  30 days post-baseline: number analyzed (Participants) | 12 | 12 | 11 | 14
  30 days post-baseline | 5 | 3 | 2 | 6
  90 days post-baseline: number analyzed (Participants) | 10 | 12 | 13 | 15
  90 days post-baseline | 6 | 5 | 3 | 7
  180 days post-baseline: number analyzed (Participants) | 9 | 8 | 11 | 11
  180 days post-baseline | 1 | 4 | 6 | 8

15. Secondary Outcome: Anxiousness as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 2-3 anxiousness at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 23 | 19 | 22 | 21
  Baseline | 7 | 7 | 7 | 7
  30 days post-baseline: number analyzed (Participants) | 12 | 11 | 11 | 14
  30 days post-baseline | 4 | 2 | 3 | 5
  90 days post-baseline: number analyzed (Participants) | 10 | 12 | 13 | 16
  90 days post-baseline | 4 | 3 | 3 | 3
  180 days post-baseline: number analyzed (Participants) | 9 | 9 | 11 | 11
  180 days post-baseline | 0 | 4 | 3 | 1

16. Secondary Outcome: Sadness as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 2-3 sadness at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 23 | 20 | 22 | 21
  Baseline | 5 | 3 | 7 | 3
  30 days post-baseline: number analyzed (Participants) | 12 | 12 | 11 | 14
  30 days post-baseline | 3 | 1 | 1 | 2
  90 days post-baseline: number analyzed (Participants) | 10 | 12 | 13 | 14
  90 days post-baseline | 4 | 4 | 2 | 2
  180 days post-baseline: number analyzed (Participants) | 9 | 8 | 12 | 10
  180 days post-baseline | 0 | 0 | 3 | 2

17. Secondary Outcome: Fatigue as Measured by the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
Description: Participants reporting Grade 2-3 fatigue at baseline and post-baseline (30 days, 90 days, and 180 days) in the HOPE RCT. {Symptoms were graded in accordance with the established composite grading algorithm, with higher grades corresponding to worse outcomes.}
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Fitbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Participants
  Baseline: number analyzed (Participants) | 22 | 18 | 21 | 22
  Baseline | 7 | 7 | 12 | 15
  30 days post-baseline: number analyzed (Participants) | 12 | 12 | 11 | 15
  30 days post-baseline | 3 | 4 | 4 | 8
  90 days post-baseline: number analyzed (Participants) | 10 | 12 | 12 | 15
  90 days post-baseline | 5 | 2 | 5 | 6
  180 days post-baseline: number analyzed (Participants) | 9 | 7 | 10 | 11
  180 days post-baseline | 2 | 0 | 4 | 5

18. Secondary Outcome: Correlation Between Patient and Physician Estimates of Performance Status as Assessed by ECOG-PS (HOPE RCT)
Description: Patients' and their physicians' ECOG-PS measurements taken at baseline and post-baseline (30 days, 90 days, and 180days) in the HOPE RCT. Weighted Kappa statistics calculated at each timepoint to assess correlation.
Time Frame: Baseline, 30 days, 90 days, 180 days (Phase II)
Population: Participants who had both physician- and patient-reported ECOG Performance Status (PS) assessed at baseline and/or follow-up timepoints.
Measure: Number; unit: Weighted Kappa (no unit)
Groups:
- Arm 2: Firbit + Passive App: Participants were asked to wear the Fitbit Charge 2. The HOPE app will also collect passive smartphone data.
Arm/Group | Arm 1: Fitbit + Active App | Arm 2: Firbit + Passive App | Arm 3: Active App | Arm 4: Passive App
Number analyzed (Participants) | 23 | 21 | 22 | 22
Weighted Kappa (no unit)
  Baseline: number analyzed (Participants) | 21 | 16 | 18 | 17
  Baseline | 0.70 | 0.48 | 0.35 | 0.39
  30 days post-baseline: number analyzed (Participants) | 18 | 19 | 19 | 18
  30 days post-baseline | 0.24 | 0.59 | 0.61 | 0.34
  90 days post-baseline: number analyzed (Participants) | 11 | 14 | 9 | 8
  90 days post-baseline | 0.20 | 0.31 | -0.15 | 0.17
  180 days post-baseline: number analyzed (Participants) | 7 | 12 | 10 | 10
  180 days post-baseline | -0.08 | 0.71 | 0.24 | 0.25

ADVERSE EVENTS:
Time Frame: HOPE Pre-Pilot: 30 days; HOPE RCT (4 arms): 180 days; SMART: 90 days
Description: Only death and serious adverse events were assessed for the SMART Study Arm.
Groups:
- HOPE Pre-Pilot: 10 patients will be enrolled in stage 1 to refine the HOPE App intervention; All participants will receive: HOPE App, The Fitbit Zip, The Fitbit Charge 2
  The amount of step collected by each device will be compared. This will allow the team to identify which wearable accelerometer to use in stage 2.
  Fitbit Zip: Fitbit Zip HOPE App: HOPE App Fitbit Charge 2: Fitbit Charge 2
Arm/Group | HOPE Pre-Pilot | Refined Smartphone App and Accelerometer (HOPE) | Wearable Accelerometer (HOPE) | Refined Smartphone App (HOPE) | Usual Care (HOPE) | SMART Study Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/23 | 0/21 | 0/22 | 2/22 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/23 | 0/21 | 0/22 | 0/22 | 0/4
Other Adverse Events (participants affected / at risk) | 10/10 | 22/23 | 19/21 | 21/22 | 18/22 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HOPE Pre-Pilot (N=10) | Refined Smartphone App and Accelerometer (HOPE) (N=23) | Wearable Accelerometer (HOPE) (N=21) | Refined Smartphone App (HOPE) (N=22) | Usual Care (HOPE) (N=22) | SMART Study Arm (N=0)
Constipation (Gastrointestinal disorders) | 4 | 10 | 11 | 10 | 10 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 5 | 5 | 4 | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 8 | 8 | 7 | 9 | 0
Vomit (Gastrointestinal disorders) | 1 | 3 | 2 | 3 | 3 | 0
Neuropathy (Nervous system disorders) | 4 | 12 | 13 | 10 | 8 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 11 | 9 | 9 | 11 | 0
Anxiety (Nervous system disorders) | 8 | 18 | 18 | 17 | 16 | 0
Depression (Nervous system disorders) | 8 | 11 | 8 | 9 | 9 | 0
Fatigue (Nervous system disorders) | 10 | 22 | 19 | 21 | 17 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT03022032/Prot_SAP_000.pdf